CLINICAL TRIAL: NCT05134285
Title: The Effects of Recurrent PE on Women and Offspring's Health
Brief Title: Effects of Recurrent PE on Women and Offspring
Acronym: RPOH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dunjin Chen (Other)
Responsible Party: Sponsor-Investigator, Dunjin Chen, Director, Guangzhou Medical University
Organization: Guangzhou Medical University (Other)
Other Study IDs: 81830045
Record Dates: First submitted 2021-11-08; First posted 2021-11-24 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Preeclampsia; Recurrence; Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Recurrence; Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: pregnancy without preeclampsia
  Interventions: Other: blood pressure,BMI, blood sample
- preeclampsia: pregnancy complicated with preeclampsia at the first delivery or at the second delivery
  Interventions: Other: blood pressure,BMI, blood sample
- recurrent preeclampsia: pregnancy complicated with preeclampsia at two deliveries
  Interventions: Other: blood pressure,BMI, blood sample

INTERVENTIONS:
Other: blood pressure,BMI, blood sample — Blood pressure will be monitored. BMI will be measured. Blood samples will be tested.

SUMMARY:
The purpose of this study is to evaluate the risk factors of recurrent preeclampsia and compare the short-term and long-term adverse outcomes of women and their offspring.

DETAILED DESCRIPTION:
The investigators collected women delivered twice in a row in our hospital. The investigators divided these pregnant women into three groups. Women in the first group did not complicate preeclampsia at both deliveries; Women in the second group complicated preeclampsia at the first delivery or at the second delivery; women in the third group complicated preeclampsia at two deliveries. The investigators explore the risk factors of recurrent preeclampsia and measure blood pressure, blood lipids, thyroid function, glycosylated hemoglobin, ALT, AST, et al. in one year, three years, and five years after the second delivery.

ELIGIBILITY:
Inclusion Criteria:

* women with at least twice of delivery history

Exclusion Criteria:

* women with chronic hypertension

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women with at least twice of delivery history are divided into three groups, control group refers to women without preeclampsia history, the second group refers to women complicated with preeclampsia at the first delivery or at the second delivery, the third group refers to women complicated with preeclampsia at two deliveries.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
blood pressure and hypertension of women | 1year after the second deliver
  blood pressure ≥140/90 mmHg
blood pressure and hypertension of women | 3 years after the second deliver
  blood pressure ≥140/90 mmHg
blood pressure and hypertension of women | 5 years after the second deliver
  blood pressure ≥140/90 mmHg
blood pressure and hypertension of offspring | 1 year old
  blood pressure≥140/90 mmHg
blood pressure and hypertension of offspring | 3 years old
  blood pressure≥140/90 mmHg
blood pressure and hypertension of offspring | 5 years old
  blood pressure≥140/90 mmHg
level of glycosylated hemoglobin in blood | 1 year after the second deliver
  women
level of glycosylated hemoglobin in blood | 3 years after the second deliver
  women
level of glycosylated hemoglobin in blood | 5 years after the second deliver
  women
level of cholesterol, LDL, HDL, VLDL-C in blood | 1 year after the second deliver
  women
level of cholesterol, LDL, HDL, VLDL-C in blood | 3 years after the second deliver
  women
level of cholesterol, LDL, HDL, VLDL-C in blood | 5 years after the second deliver
  women
level of FT3,FT4, and hTSH in blood | 1year after the second deliver
  women
level of FT3,FT4, and hTSH in blood | 3 years after the second deliver
  women
level of FT3,FT4, and hTSH in blood | 5 years after the second deliver
  women
level of AST and ALT in blood | 1year after the second deliver
  women
level of AST and ALT in blood | 3 years after the second deliver
  women
level of AST and ALT in blood | 5 years after the second deliver
  women

SECONDARY OUTCOMES:
BMI of offspring | 1 year old
  weight(kg)/height(m)2
BMI of offspring | 3 years old
  weight(kg)/height(m)2
BMI of offspring | 5 years old
  weight(kg)/height(m)2
level of insulin in blood | 1year after the second deliver
  women
level of insulin in blood | 3 years after the second deliver
  women
level of insulin in blood | 5 years after the second deliver
  women
level of fructosamine in blood | 1year after the second deliver
  women
level of fructosamine in blood | 3 years after the second deliver
  women
level of fructosamine in blood | 5 years after the second deliver
  women
level of AI37℃、AI4℃、PRA、ALD、AngII in blood | 1 year after the second deliver
  women
level of AI37℃、AI4℃、PRA、ALD、AngII in blood | 3 years after the second deliver
  women
level of AI37℃、AI4℃、PRA、ALD、AngII in blood | 5 years after the second deliver
  women

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Key Laboratory for Major Obstetric Diseases of Guangdong Province, The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No